CLINICAL TRIAL: NCT03912779
Title: The Role of Interactive Hearing Aid Self-management Education on Self-efficacy for Hearing Aid(s), Readiness for Action and Hearing Aid Knowledge in First Time Hearing Aid Users
Brief Title: Evaluation of Self-management Education in First Time Hearing Aid Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Aston University (Other)
Responsible Party: Principal Investigator, Melanie Ferguson, Associate Professor, Study Principal Investigator, Nottingham University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16IH006; 168-2016-RGM (Other: Aston University)
Record Dates: First submitted 2019-02-22; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Hearing Loss
Keywords: First time hearing aid user
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C2Hear RLOs (Experimental): C2Hear RLOs (https://www.youtube.com/C2HearOnline): nine (custom earmould) or eight (open fit hearing aid) multi-media learning clips covering practical and psychosocial components of owning a hearing aid, alongside user testimonials (n= 7). Participants asked to watch all relevant to their prospective hearing aid coupling (custom earmould or open fit), with no limit on number of views. A paper diary documented usage during the study duration.
  Interventions: Behavioral: C2Hear RLOs
- Printed hearing aid booklet (Placebo Comparator): A 32-page printed A5 colour booklet, designed and written by local Audiology staff, supplied to all prospective hearing aid owners at the study centre as standard care. Same booklet supplied irrespective of hearing aid style (custom/open fit). All content conveyed via text and supporting pictures only. Participants assigned to the placebo comparator were asked to read the booklet once. A paper diary documented usage during the study duration.
  Interventions: Behavioral: Printed hearing aid booklet

INTERVENTIONS:
Behavioral: C2Hear RLOs — Freely available online RLOs
  Arms: C2Hear RLOs
Behavioral: Printed hearing aid booklet — Departmental printed hearing aid booklet (standard care)
  Arms: Printed hearing aid booklet

SUMMARY:
The study will assess the impact of a hearing aid self-management intervention in first time hearing aid users compared to standard hearing aid self-management. Namely, the C2Hear multimedia videos, or Reusable Learning Objects (RLOs) will be used as the self-management intervention. A departmental hearing aid booklet (standard clinical care) will be used as the control intervention.

The study will determine the role of these RLOs in self-efficacy for hearing aid(s), hearing aid knowledge and readiness for action compared with standard hearing aid self-management education (hearing aid booklet) in groups of first time hearing aid users. Both groups will receive the education at the earliest audiology appointment (hearing assessment), helping to distinguish any impact of earlier education delivery.

DETAILED DESCRIPTION:
Research question: To assess the role of interactive hearing aid self-management education on self-efficacy for hearing aid(s), readiness for action and hearing aid knowledge in first time hearing aid users.

Objectives:

Primary research question:

- Does the early delivery of interactive hearing aid self-management education improve self-efficacy for hearing aid(s) compared with standard care in first-time hearing aid users?

Secondary research questions:

i. Does the early delivery of interactive hearing aid self-management education improve readiness for hearing aids (their chosen intervention) compared with standard care in first-time hearing aid users?

ii. Does the early delivery of interactive hearing aid education improve hearing aid knowledge compared with standard care in first-time hearing aid users?

Study design:

A single centre, prospective study with two randomised arms; intervention group (access to RLOs in DVD/ or online format, patients' preference) and control (standard hearing aid education booklet).

Prospective first-time hearing aid users will be invited to take part in the study at hearing assessment, where they will be randomised to either the control or intervention group. Following 6-8 weeks of independent use prior to receiving hearing aids, study investigators will assess the impact of each education type on individuals self-efficacy for hearing aids, readiness for action and hearing aid knowledge.

Comparisons will be made to previous evaluation of the RLOs to allow exploration of the impact of earlier hearing aid self-management education on self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years
* Prospective first-time hearing aid users (defined as no hearing aid use in the last 2 years)
* English as their spoken language or good understanding of English

Exclusion Criteria:

* Those unable to complete study questionnaires due to age-related problems (e.g. cognitive decline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Measure of Audiologic Rehabilitation Self-efficacy for Hearing Aids score (West and Smith, 2007) | Change from Baseline self-efficacy for hearing aids up to 8 weeks
  Self-reported self-efficacy for hearing aid(s) measured across four-subscales (Basic/advanced handling, adjustment to hearing aids and aided listening). Participants rank confidence in the tasks/behaviours described using an 11-point scale (0%=cannot do this, to 100%=certain I can do this).

SECONDARY OUTCOMES:
Hearing aid self-efficacy using Ida Motivational Line Tools (Ida Institute, 2013) | Change from Baseline self-efficacy for hearing aids up to 8 weeks
  Self-report hearing aid self-efficacy (Ida Line Tool Question 2) determines participants perceived confidence in their ability to use hearing aid(s) using an 11-point visual analogue scale (0 = not at all confident, to 10= very much confident).
Hearing Aid and Communication Knowledge (HACK: Ferguson et al., 2015) | Up to 8 weeks
  A 20-item open-ended questionnaire that measures free recall of hearing aid knowledge relevant to practical (n = 12) and psychosocial (n = 8) issues on hearing aids and communication. One point is allocated to each correct response, resulting in a percentage correct for each score. Maximum correct scores are 54; 32 points for practical subscale and 22 points for psychosocial subscale. Higher percentage values represent better knowledge.
Readiness for hearing rehabilitation (action); Ida Motivational Line Tools Question 1 (Ida Institute, 2013) | Change from Baseline readiness up to 8 weeks
  Self-report readiness for hearing rehabilitation (action) (Ida Line Tool Question 1) determines participants readiness to use hearing aid(s) using an 11-point visual analogue (0 = not at all important, to 10= very much important).

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Ferguson, Principal Investigator — Nottingham University Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No